CLINICAL TRIAL: NCT03099746
Title: A Clinical Trial of Decision Support for End of Life Care Among Surrogate Decision Makers of the Chronically Critically Ill
Brief Title: Decision Support Among Surrogate Decision Makers of the Chronically Critically Ill (INVOLVE)
Acronym: INVOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ronald Hickman, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08-16-25; 5R01NR015750-02 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-04-04 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Critical Illness
Keywords: chronically critically ill; surrogate decision maker
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- INVOLVE (Experimental): The first study condition, called "Interactive Virtual Decision Support for End-of-Life and Palliative Care (INVOLVE)" will consist of exposures to an avatar-based decision support technology that will be administered via tablet computer and allow SDMs opportunities to practice their communication and decision making skills through interactions with avatars that portray a decision coach and various healthcare providers.
  Interventions: Behavioral: INVOLVE
- Informational Support (Experimental): The second condition, called Informational Support (IS), will also be administered via tablet computers and expose SDMs to educational resources of INVOLVE without the experiential components.
  Interventions: Behavioral: Informational Support
- Usual Care (Experimental): The third condition, usual care (UC), will expose SDMs to the routine communication and decisional support practices provided by the healthcare team.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: INVOLVE — Interactive content and decision coaching with tailored framing of messages to subject's informational processing style and stage of change to promote participatory decision making behavior. Consideration of options, consequences, values, and preferences to formulate an informed decision.
  Arms: INVOLVE
Behavioral: Informational Support — Passive, non-tailored informational support. Screen-based education (videos) with information content on advance care decisions that occur in the intensive care unit.
  Arms: Informational Support
Behavioral: Usual Care — Routine decision support practices by the healthcare team. Family meetings, bedside updates, and access to printed or electronic decision aids.
  Arms: Usual Care

SUMMARY:
Each year, millions of Americans are admitted to an intensive care unit (ICU). For more than half of them, ICU admission initiates a cascade of decisions about treatment and end-of-life care.This is particularly the case for patients with chronic critical illness, a life-limiting syndrome. Most (74%-82%) ICU patients who require mechanical ventilation have transient or persistent cognitive impairment that precludes them from making their own healthcare decisions. Among ICU patients, the chronically critically ill (CCI) are at highest risk for cognitive impairment and thus require a surrogate decision maker (SDM), usually a family member. SDMs for the critically ill often describe high states of psychological stress associated with the uncertainty of the patient's condition and their decision making role.

The purpose of this study is to test the effectiveness of two decision support interventions for end-of-life care delivered to SDMs of CCI patients. This will be the first study to test interventions tailored to the unique needs of the SDMs of CCI patients delivered using an interactive avatar based format.

DETAILED DESCRIPTION:
The investigators will conduct a three-arm unblinded clinical trial using pre- and post-tests to evaluate the efficacy of two electronic decision-support interventions, Interactive Virtual Decision Support for End-of-Life and Palliative Care (INVOLVE) and Informational Support (IS), compared to each other and to usual care (UC) among 270 SDMs of cognitively impaired CCI patients. This design will allow the investigators to prospectively compare the efficacy of the experiential avatar-based decision support tool (INVOLVE) with both an information-only condition and UC. Subjects assigned to an experimental condition (INVOLVE or IS) will receive two doses of the intervention, at enrollment and 1 day later. After the second dose, these subjects will have access to their assigned condition for subsequent self-administered doses, which will be electronically captured until the patient's ICU discharge or death. Data will be collected at (T1) baseline (Day 3 or 4 of the patient's ICU stay), and then on Days 1, 3, 7 and 90 post-baseline

.

The investigators aim to:

1. Identify the essential elements of the graphical user interface and educational content needed to revise the INVOLVE prototype for a set of common end-of-life decisions that occur in the ICU.
2. Evaluate if there are differences in the decision making readiness and decision making quality between subjects exposed to INVOLVE, IS, or UC on Days 1, 3, and 7 days post-baseline while accounting for covariates (prior SDM experience, SDM knowledge of the patient's preferences, and SDM's religious beliefs).
3. Determine if there are differences in the post-decision outcomes of SDMs and their CCI patient by study condition while accounting for covariates at 90 days post-baseline.

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for CCI patients:

* aged 18 years or older
* required mechanical ventilation and ICU stay for greater than or equal to 3 days
* not expected to be transferred out of the ICU within 48 hours
* lacks cognitive capacity, as determined by a Glasgow Coma Scale eye score of less than 3 or the motor score less than 6 and verifying the status by asking the patients's attending physician or advanced practice nurse whether he or she would obtain consent from the patient or a family member
* has an identified SDM (next-of-kin or legal representative for healthcare decision making).

Eligibility criteria for SDMs:

* aged 18 years or older
* identified by the healthcare team as the patient's next of kin or legal representative for healthcare decision making
* able to speak and understand English
* able to view images on an 10-inch computer screen and hear audio through a standard set of headphones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Repeated Measures | From (T1) baseline through (T5) 90 days post-baseline
  ANOVA Model (F-Statistic)

SECONDARY OUTCOMES:
Change in Preparation for Decision Making Scale | (T1) baseline through (T4) 7 days post-baseline
  Measure of Decision Making Preparedness
Change in Family Decision Making Self-Efficacy Scale | (T1) baseline through (T4) 7 days post-baseline
  Measure of Decision Making Self-Efficacy
Change in Single item measure of Role Stress | (T1) baseline through (T4) 7 days post-baseline
  Measure of Decisional Role Stress
Change in Decision Conflict Scale | (T1) baseline through (T4) 7 days post-baseline
  Measure of Decision Conflict
Change in Modified Control Preferences Scale | (T1) baseline through (T4) 7 days post-baseline
  Measure of Behavioral Activation
Change in Decision Regret Scale | (T1) baseline and (T5) 90 days post-baseline
  Measure of Decision Regret
Change in Hospital Anxiety and Depression Scale | (T1) baseline and (T5) 90 days post-baseline
  Measure of Anxiety and Depressive Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ronald L. Hickman, PhD, RN, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pignatiello GA, Tuschman PJ, Griggs S, Schiltz NK, Hoffer A, Hickman RL Jr. Rethinking Regret: Reappraisal Tendencies Buffer Regret for ICU Surrogates Following Patient Death. West J Nurs Res. 2025 Sep;47(9):799-809. doi: 10.1177/01939459251344205. Epub 2025 Jun 16. PMID 40521758
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350